CLINICAL TRIAL: NCT04881981
Title: INT-SCART-001: A Phase I Study Evaluating the Safety of Stereotactic Central Ablative Radiation Therapy (SCART) for Bulky Metastatic or Recurrent Cancer.
Brief Title: A Phase I Study Evaluating the Safety of Stereotactic Central Ablative Radiation Therapy (SCART) for Bulky Metastatic or Recurrent Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Baptist Health, Louisville (Other)
Collaborators: Drexel University (Other); Innovative Institute (Unknown); University of Kentucky (Other); Foshan Chancheng Hospital (Unknown)
Responsible Party: Principal Investigator, Weisi Yan, Medical Director, Baptist Corbin Radiation Oncology, Baptist Health, Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT-SCART-001
Record Dates: First submitted 2021-05-06; First posted 2021-05-11 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Malignant Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: 3+3 phase one trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- SCART Arm (Experimental): Single Arm patients will be treated with SCART to different dose levels.
  Interventions: Radiation: SCART radiation therapy

INTERVENTIONS:
Radiation: SCART radiation therapy — We will deliver high dose radiation therapy using SCART method. Beam energies of 6Mv will be used. The high dose SCART therapy will be delivered using LINAC systems, as available and appropriate for each patient. The treatment plan used for each patient will be based on an analysis of the volumetric dose including DVH analyses of the PTV and critical normal structures.

SUMMARY:
We aim to evaluate the feasibility and toxicity of testing the tolerance and immunogenic effects of high-dose SCART radiotherapy in patients with bulky metastatic or recurrent cancer in the setting of a single-arm phase I clinical trial.

The primary endpoint of the study was to determine dose-limiting toxicities (DLT)s and the Maximum Tolerated Dose (MTD) of SCART to bulky metastatic or recurrent cancers.

DETAILED DESCRIPTION:
Despite advances in screening and surveillance, patients continue to present with both bulky primary and metastatic tumors. Some patients presented with recurrent bulky cancer in prior treated radiation fields. Spatially Fractionated Radiation therapy (SFRT) has a history of over 100 years. The principle of SFRT is distinctive from the standard radiation approaches, as it treats the total tumor with a non-uniform dose, effectively treating the tumor while staying within normal tissue tolerance of the surrounding structures. Historically, SFRT is frequently used to treat bulky malignant tumors with a high radiation dose in the stereotactic radiosurgery (SRS)/stereotactic body radiotherapy (SBRT) dose range (10-20 Gy per fraction) using megavoltage x-ray beams. The application of SFRT, historically known as GRID therapy, has produced dramatic relief of severe symptoms, significant objective regression, above average local control rates and minimal toxicity in palliative settings.

High-dose GRID radiotherapy, sometimes termed spatially-fractionated GRID radiotherapy (SFGRT), is a treatment modality that was introduced in 1909 and commonly used through the 1930's . In 1909, Kohler in Germany described radiation delivered through a perforated screen with regularly spaced blocked areas that created an effect similar to treatment with multiple small pencil beams. This spatially fractionated radiation, in contradistinction to current approaches, does not attempt to treat the total tumor volume with a uniform dose. Instead, this technique allows the delivery of high doses of radiation in clusters of small areas without producing prohibitive normal tissue damage to skin and subcutaneous tissues. In its early applications, two-dimensional grid fields were used, typically with orthovoltage beams. The grids were usually composed of open/shield circular or square shapes ranging in size from 0.5 to 1.5 cm. The application was mainly for the treatment of advanced bulky tumors.

However, the technique of GRID radiotherapy has not evolved significantly since its inception in the early 1900's, and is not the optimal method of delivering spatially fractionated radiation in the modern era. GRID has the limitation of delivering relatively high doses of radiation to normal tissues, depending on tumor location, as it is delivered via a single beam that must pass through normal tissues to reach its target. Most importantly, the highest-dose regions of the grid are superficial, and often are outside of the tumor target itself.

The basic principle of the LATTICE Radiotherapy (LRT) is to create within tumor volume multiple localized high-dose islands (12 Gy and higher) with a certain degree of separation to form low dose regions (3 Gy or lower). In an extreme case, one or two focused dose islands could be introduced in a small tumor.

Modern radiotherapy methods are readily available to deliver 3D high-dose LATTICE radiotherapy with superior dosimetry compared to the 2D GRID technique . An array of focused high-dose volumes, in essence a lattice of doses in 3D, can be generated through modern techniques resulting in highly heterogeneous dose distributions within the tumor volume, leaving adjacent and peripheral normal tissue minimally exposed.

Similar to the core principles and concepts of LRT, SCART aims to stereotactically irradiate part of target volume (hotspot) located at the center of a large tumor target with an ablative dose (15Gy or higher) and the dose quickly falls off from the edge of hotspot to low dose (3Gy or lower) at the edge of tumor volume. The goal is to irradiate as large a volume as possible with ablative dose, while maintaining the dose to the border of the tumor at low dose.

SCART is a different approach which pursuits not only the dose escalation but also the idea of facilitating or promoting intra-tumoral bystander effect, thus increasing the biological effectiveness of the treatment. Published data reviewed by Peters, et al. strongly suggest that GRID therapy induces a rapid and higher rate of tumor cell apoptosis in bulky and hypoxic tumors. This technique is very appealing to treat patients with voluminous gynecological tumors.

These makes SCART Radiotherapy a practically achievable alternative to traditional GRID therapy and LATTICE, which delivers a highly heterogeneous dose distribution, anticipated to trigger the bystander effect of radiation. With high dose regions strictly contained within the target volume, normal tissue toxicity is practically avoided providing an increased therapeutic ratio.

SCART is a promising tool to achieve dose escalation which will lead to a higher local control without adding any extra toxicity in the peripheral normal tissue regions.

ELIGIBILITY:
Inclusion Criteria:

3.1.1 Patients must have a history of histologically confirmed metastatic or recurrent cancers.

3.1.2 Patients must have measurable disease documented by CT and/or PET that is amenable for SCART radiation with the shortest axis of 3 cm or longer.

3.1.3 Patients must be 18 years of age or older, as this is not a pediatric protocol. There is no maximum age restriction.

3.1.4 Patients must have a life expectancy of at least 6 months in order for the study endpoints to be evaluable.

3.1.5 Patients must have a Zubrod/GOG performance status of 0 or 1.

3.1.6 Patients must have normal organ and marrow function as defined below: leukocyte>3,000/m l absolute neutrophil count >1,500/m l platelets >100,000/m l bilirubin within normal institutional limits AST(SGOT)/ALT(SGPT) 2.5 X institutional upper limit of normal Creatinine within normal institutional limits OR; Creatinine clearance > 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.

3.1.7 Women of child-bearing potential will be asked to use adequate contraception.

3.1.8 Patients must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

3.2.1 Women who are pregnant or breastfeeding will be excluded.

3.2.2 Patients must not have any co-morbidity with life expectancy ≤ 6 months, or any uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

3.2.3 Patients must not have active Crohn's disease or inflammatory bowel disease (IBD).

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-06-05 (Estimated); Primary Completion 2022-05-05 (Estimated); Study Completion 2022-05-05 (Estimated)

PRIMARY OUTCOMES:
Toxicity | 12 months
  radiation treatment-related grade 3+ non-hematologic adverse events

SECONDARY OUTCOMES:
Assessment of the antitumor effect | 12 months
  PR or CR defined by radiology.
Evaluation of quality of life (QoL). | 12 months
  Evaluation of quality of life (QoL).
Biomarkers | 3-6 months
  T cell activities and/or NGS sequencing

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - Innovative Cancer Institute, Miami, Florida
  - Baptist health, Corbin, Kentucky
  - University of Kentucky Morehead Cancer Treatment Center, Morehead, Kentucky
- Foshan Chancheng Hospital, Foshan, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Physics plans and DVHs. Biomarker data from patients treated with SCART.
Supporting Information: Study Protocol, CSR
Time Frame: 1 year after the publication and for 5 years.

REFERENCES:
- [Background] Yan W, Khan MK, Wu X, Simone CB 2nd, Fan J, Gressen E, Zhang X, Limoli CL, Bahig H, Tubin S, Mourad WF. Spatially fractionated radiation therapy: History, present and the future. Clin Transl Radiat Oncol. 2019 Oct 22;20:30-38. doi: 10.1016/j.ctro.2019.10.004. eCollection 2020 Jan. No abstract available. PMID 31768424
- [Background] Jiang L, Li X, Zhang J, Li W, Dong F, Chen C, Lin Q, Zhang C, Zheng F, Yan W, Zheng Y, Wu X, Xu B. Combined High-Dose LATTICE Radiation Therapy and Immune Checkpoint Blockade for Advanced Bulky Tumors: The Concept and a Case Report. Front Oncol. 2021 Feb 12;10:548132. doi: 10.3389/fonc.2020.548132. eCollection 2020. PMID 33643893
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6872856/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/33643893/